CLINICAL TRIAL: NCT01461694
Title: Comparison of Intense Pulsed Light System 650 Advance Hand-Piece and Alexandrite Laser for Female Facial Hair Reduction
Brief Title: Facial Hair Reduction Using Intense Pulsed Light (IPL) & Alexandrite Laser
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: NHS Greater Glasgow and Clyde (Other)
Responsible Party: Principal Investigator, Adam Gilmour, Clinical Laser Research Fellow, NHS Greater Glasgow and Clyde
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GN11SU380
Record Dates: First submitted 2011-10-25; First posted 2011-10-28 (Estimated); Last update posted 2012-05-14 (Estimated); Status verified 2012-05

CONDITIONS: Hirsutism
Keywords: Hirsutism; Laser; Hair Reduction; IPL; Intense Pulsed Light
MeSH Terms: conditions — Hirsutism | interventions — Intense Pulsed Light Therapy; Lasers, Solid-State

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- IPL (Active Comparator): Half face treated with IPL
  Interventions: Device: Intense Pulsed Light (IPL)
- Alexandrite Laser (Active Comparator): Half face treated with Alexandrite Laser
  Interventions: Device: Alexandrite Laser

INTERVENTIONS:
Device: Intense Pulsed Light (IPL) — Half Face Treated with IPL
  Arms: IPL
Device: Alexandrite Laser — Half face treated with Alexandrite Laser
  Arms: Alexandrite Laser

SUMMARY:
The purpose of this study is to compare the efficacy of the IPL system 650advance handpiece with the alexandrite laser for the purposes of female facial hair reduction

DETAILED DESCRIPTION:
This is a randomised (splitface)controlled trial, comparing the use of the Intense Pulsed Light (IPL) system 650 advance handpiece against the Alexandrite Laser for the purposes of female facial hair reduction. Previous studies have shown that the alexandrite laser is superior to IPL in achieving hair reduction. A new handpiece (Lynton, Lumina 650 advance) available for the IPL system is designed to further optimise its use in removing female facial hair (particularly those hair colours previously unresponsive to treatment). This study will compare the alexandrite laser to the IPL system using the new handpiece. This may lead to improvements in the treatment of female patients with male pattern facial hair. Female patients referred to our facial hair reduction service will be recruited to this study. 1/2 their face will be treated with IPL and 1/2 with alexandrite laser. Each participant will receive 6 full treatments at approximately 6 weekly intervals. Participants will be asked to fill in a satisfaction questionnaire and have clinical photographs taken pre treatment and at 1 and 3months post final treatment. All treatments will be carried out in our dedicated laser suite at Glasgow Royal Infirmary.

ELIGIBILITY:
Inclusion Criteria:

* Female Patients
* Minimum age 16years old
* Fitzpatrick skin types I-III
* Significant facial hair.

Exclusion Criteria:

* Fitzpatrick skin types IV-VI
* Age less than 16years old
* Males
* No visible facial hair growth
* Use of electrolysis or depilatory creams 6weeks prior to treatment
* Active acnes
* Current coldsore
* Previous facial hair removal with laser or IPL in past 12 months
* Sun tanned skin

Min Age: 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2011-11; Primary Completion 2013-03 (Estimated); Study Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
Change in total Hair Count measurement at 1month post final treatment from baseline | Baseline and 1 month
  Pre Treatment hair count assessed using videomicroscopy as baseline. Post final treatment hair counts will be measured again at 1month to assess if there has been a reduction in total hair count from pre-treatment
Change in total hair count at 3months post final treatment from baseline | Baseline and 3months post final treatment
  Pre Treatment hair count assessed using videomicroscopy as baseline. Post final treatment hair counts will be measured again at 3months to assess if there has been a reduction in total hair count from pre-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Adam Gilmour, MBChB, MRCS (Ed), Principal Investigator — NHS Greater Glasgow & Clyde; Iain Mackay, MBChb, MRCS, FRCS (plast), Study Chair — NHS Greater Glasgow & Clyde; Vivek Sivarajan, MBChB, MRCS, MD, FRCS (Plas), Study Director — NHS Greater Glasgow & Clyde
Locations (1):
- Canniesburn Plastic Surgery Unit, Glasgow Royal Infirmary, Glasgow, United Kingdom